CLINICAL TRIAL: NCT03370068
Title: The Role of Intracytoplasmic Sperm Injection in Non-male Factor Infertility in Maternal Age Above 39
Brief Title: The Role of ICSI in Non-male Factor Infertility in Advanced Maternal Age
Acronym: ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Tal Miller-Elkan (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Tal Miller-Elkan, Principal Investigator, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SHEBA-17-4531-TEM-CTIL
Record Dates: First submitted 2017-11-20; First posted 2017-12-12 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Infertility, Female
Keywords: ICSI; IVF; Infertility; non-male factor; intracytoplasmic sperm injection; In vitro fertilization
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI (Experimental): All the oocytes in this group (from one ovary) will undergo insemination by ICSI.
  Interventions: Other: ICSI
- Conventional IVF (Active Comparator): All the oocytes in this group (from the other ovary) will undergo insemination by conventional IVF.
  Interventions: Other: Conventional IVF

INTERVENTIONS:
Other: ICSI — Oocytes retrieved from one ovary will undergo insemination by ICSI.
  Arms: ICSI
Other: Conventional IVF — Oocytes retrieved from the second ovary will undergo insemination by conventional IVF
  Arms: Conventional IVF

SUMMARY:
The use of Intracytoplasmic sperm injection (ICSI) has increased in the last decades regardless of the cause of infertility. Despite the increased use there is no clear evidence that ICIS is more effective than conventional in vitro fertilization (IVF) for non-male factor infertility. The investigators therefore aim to perform a prospective randomized controlled study to compare between ICSI and conventional IVF in women between 39 to 44 years of age with non-male factor infertility.

DETAILED DESCRIPTION:
ICSI is a method used in IVF in which a single sperm is injected directly into an oocyte. Originally ICSI was developed as a method for the treatment for couples with severe male factor infertility. In the last decades the use of ICSI has increased dramatically, especially for non-male factor infertility. In certain fertility clinics in the world ICSI is conducted in 100% of IVF cycles.

Despite the increased use of ICSI, there is no clear evidence that ICIS is more effective than conventional IVF for non-male factor infertility. There are currently few randomized controlled studies that compared the two modalities in the case of non-male factor infertility. In a randomized controlled trial that included 415 couples with non-male factor infertility and women younger than 37 years of age, conventional IVF was associated with better fertilization and implantation rates than ICSI but with comparable live birth rates. In addition, studies have not shown an advantage for ICSI over conventional IVF in the case of unexplained infertility, low oocyte yield or routine use to decrease the incidence of fertilization failure.

The proportion of women after the age of 35 undergoing IVF is constantly on the rise. Oocytes retrieved from older women are often of lower quality then oocytes retrieved from younger women. It is believed that due to the lower quality the fertilization rate is decreased in this population. However a recently published retrospective study including 745 women did not show an advantage for ICSI over conventional IVF. Contrary to what is believed, the conventional IVF group had a higher number of zygotes formed, more cycles with embryos transferred at the blastocyst stage and more cycles where embryos were available for cryopreservation.

The investigators therefore aim to perform a prospective randomized controlled study to compare between ICSI and conventional IVF in women between 39 to 44 years of age with non-male factor infertility. Male-factor infertility will be diagnosed according to the accepted semen analysis values included a semen concentration of 200 million/mL, progressive motility of 40% and a strict morphology of 4%. Patients will undergo standard clinical and hormonal investigation as usual for IVF. The treatment protocol will be in accordance with the decision of the attending physician, regardless of the research. Randomization will be between the ovaries of each patient. Following an informed consent a computer based randomization will allocate either ICSI or conventional IVF for each ovary so that for each study participant oocyte from one ovary will be randomly allocated to insemination by ICSI and the oocytes from the other ovary will be allocated to insemination by conventional IVF. As is customary in our IVF unit, 24, 72 and 96 hours after oocyte retrieval, the embryos will by studied by an embryologist for the number of cells and embryo quality.

ELIGIBILITY:
Inclusion Criteria:

* Women between 39 to 44 years of age undergoing IVF treatments for non-male factor infertility.

Exclusion Criteria:

* Women undergoing IVF treatments for male factor infertility.
* Cases where PGD is planned.
* Women with a BMI above 40.
* Women younger then 39 years of age or older then 44 years of age.
* Women with a rate of fertilization bellow 50% in previous IVF cycles.

Ages: 39 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | 1 day
  The rate of fertilized oocytes

SECONDARY OUTCOMES:
Embryos | 3-4 day
  Number of embryos day 2/3
Top quality embryos | 3-4 days
  Number of top quality embryos day 2/3. Embryos will be defined as top quality if they will have four cells on Day 2 and/or 7 or 8 cells on Day 3, contain <20% fragmentation, and exhibited no apparent morphological abnormalities.
Pregnancy | Approximately 2 weeks
  Pregnancy is defined as positive βhCG blood test 11-14 days after embryo transfer.
Clinical pregnancy | Approximately 6 weeks
  Clinical pregnancy is defined as gestational sac seen on vaginal ultrasound scan by 6 weeks gestation.
Pregnancy above 8 weeks gestation | Approximately 8 weeks
  Pregnancy above 8 weeks gestation with the appreance of a fetal pulse

CONTACTS AND LOCATIONS:
Overall Officials: Tal TE Elkan Miller, MD PhD, Principal Investigator — Sheba Medical Cente
Locations (1):
- IVF Unit, Sheba medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palermo G, Joris H, Devroey P, Van Steirteghem AC. Pregnancies after intracytoplasmic injection of single spermatozoon into an oocyte. Lancet. 1992 Jul 4;340(8810):17-8. doi: 10.1016/0140-6736(92)92425-f. PMID 1351601
- [Background] Boulet SL, Mehta A, Kissin DM, Warner L, Kawwass JF, Jamieson DJ. Trends in use of and reproductive outcomes associated with intracytoplasmic sperm injection. JAMA. 2015 Jan 20;313(3):255-63. doi: 10.1001/jama.2014.17985. PMID 25602996
- [Background] Bhattacharya S, Hamilton MP, Shaaban M, Khalaf Y, Seddler M, Ghobara T, Braude P, Kennedy R, Rutherford A, Hartshorne G, Templeton A. Conventional in-vitro fertilisation versus intracytoplasmic sperm injection for the treatment of non-male-factor infertility: a randomised controlled trial. Lancet. 2001 Jun 30;357(9274):2075-9. doi: 10.1016/s0140-6736(00)05179-5. PMID 11445099
- [Background] Check JH, Yuan W, Garberi-Levito MC, Swenson K, McMonagle K. Effect of method of oocyte fertilization on fertilization, pregnancy and implantation rates in women with unexplained infertility. Clin Exp Obstet Gynecol. 2011;38(3):203-5. PMID 21995144
- [Background] Luna M, Bigelow C, Duke M, Ruman J, Sandler B, Grunfeld L, Copperman AB. Should ICSI be recommended routinely in patients with four or fewer oocytes retrieved? J Assist Reprod Genet. 2011 Sep;28(10):911-5. doi: 10.1007/s10815-011-9614-9. Epub 2011 Jul 27. PMID 21792665
- [Background] Fishel S, Aslam I, Lisi F, Rinaldi L, Timson J, Jacobson M, Gobetz L, Green S, Campbell A, Lisi R. Should ICSI be the treatment of choice for all cases of in-vitro conception? Hum Reprod. 2000 Jun;15(6):1278-83. doi: 10.1093/humrep/15.6.1278. PMID 10831555
- [Background] Korkmaz C, Tekin YB, Sakinci M, Ercan CM. Effects of maternal ageing on ICSI outcomes and embryo development in relation to oocytes morphological characteristics of birefringent structures. Zygote. 2015 Aug;23(4):550-5. doi: 10.1017/S0967199414000197. Epub 2014 May 29. PMID 24869767
- [Background] Tannus S, Son WY, Gilman A, Younes G, Shavit T, Dahan MH. The role of intracytoplasmic sperm injection in non-male factor infertility in advanced maternal age. Hum Reprod. 2017 Jan;32(1):119-124. doi: 10.1093/humrep/dew298. Epub 2016 Nov 16. PMID 27852688
- [Derived] Haas J, Miller TE, Nahum R, Aizer A, Kirshenbaum M, Zilberberg E, Lebovitz O, Orvieto R. The role of ICSI vs. conventional IVF for patients with advanced maternal age-a randomized controlled trial. J Assist Reprod Genet. 2021 Jan;38(1):95-100. doi: 10.1007/s10815-020-01990-5. Epub 2020 Oct 28. PMID 33118102